CLINICAL TRIAL: NCT06081985
Title: Efficacy of Deep Transcranial Magnetic Stimulation in Patients With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bengü Yücens, Medical Doctor, Associate Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021TIPF026
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorder
Keywords: Transcranial Magnetic Stimulation; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS (Active Comparator): Deep TMS to the left dorsolateral prefrontal cortex with double-cone coil
  Interventions: Device: Transcranial Magnetic Stimulation with double-cone coil
- Sham TMS (Sham Comparator): Sham TMS to the left dorsolateral prefrontal cortex with sham coil
  Interventions: Device: Transcranial Magnetic Stimulation with sham coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation with double-cone coil — Deep Transcranial Magnetic Stimulation to the Left Dorsolateral Prefrontal Cortex with double-cone coil
  Arms: Active TMS
Device: Transcranial Magnetic Stimulation with sham coil — Transcranial Magnetic Stimulation to the Left Dorsolateral Prefrontal Cortex with sham coil
  Arms: Sham TMS

SUMMARY:
Deep TMS to the left dorsolateral prefrontal cortex intervention to reduce craving and recurrent opioid use among patients with opioid use disorder who are abstinent for at least one week.

DETAILED DESCRIPTION:
The participants will undergo baseline assessments, including rating scales and urine opioid metabolite tests. The participants will receive one of two treatments: High-frequency (10Hz, 3000 pulses per session) dTMS using a double cone coil targeting the left dorsolateral prefrontal cortex or sham stimulation. Each treatment will be preceded by a short-guided imagery (2-3 min) design to activate the relevant brain circuitry (provocation of symptoms may increase the response rate to deep TMS as was evident in the treatment of PTSD, cigarette smoking, and OCD). dTMS sessions will be conducted 10 times per week for 2 weeks, for 20 sessions. 8 weeks of patient follow-up, including clinical visits at weeks 0, 2, and 8. During this phase, subjective and objective measures of opioid use (self-report and analysis of urine samples for opioid metabolite) will be collected. Following the completion of the main part by the individual, an "open-label" treatment using the same parameters of the experiment will be offered (regardless of the treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65
* Clinical diagnosis of opioid use disorder

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Mental retardation, bipolar disorder, any psychotic disorder
* Neurological diseases such as epilepsy, ischemic stroke, multiple sclerosis
* History of head trauma that resulted in loss of consciousness for ≥5 minutes and retrograde amnesia for ≥30 minutes (self-reported history)
* Any history of seizures other than febrile childhood seizures (self-reported history)
* Clinically significant hearing impairment
* Having any prosthesis, such as an implant and pacemaker.
* Illiteracy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
craving | pretreatment, 2 weeks, and 8 weeks
  craving severity for drug use- Visual Analog Scale (VAS). The minimum and maximum values are 0-10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Impulsivity severity | pretreatment, 2 weeks, and 8 weeks
  The Barratt Impulsiveness Scale-11 (BIS). The minimum and maximum scores are 30-120. Higher scores mean a worse outcome.
Depression severity | pretreatment, 2 weeks, and 8 weeks
  The Hamilton Depression Rating Scale. The minimum and maximum scores are 0-52. Higher scores mean a worse outcome.
Anxiety severity | pretreatment, 2 weeks, and 8 weeks
  Hamilton Anxiety Rating Scale. The minimum and maximum scores are 0-56. Higher scores mean a worse outcome.
Opioid use | 8 weeks of treatment
  opioid metabolite in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Bengu Yucens, Study Director — Pamukkale University Faculty of Medicine
Locations (1):
- Bengu Yucens, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guldas S, Tumkaya S, Yucens B. Deep Transcranial Magnetic Stimulation in Patients With Opioid Use Disorder: A Double-Blind, Placebo-Controlled Randomized Trial. Addict Biol. 2025 Jun;30(6):e70057. doi: 10.1111/adb.70057. PMID 40536869